CLINICAL TRIAL: NCT05658757
Title: A Randomized Crossover Pilot Study Investigating the Impact of a "Natural" Low-Calorie Sweetener (Allulose) on Glycemic and Metabolic Measures
Brief Title: Preliminary Effect of Food Processing and Sweeteners on Glycemic and Metabolic Measures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Andrew Odegaard, Associate Professor, University of California, Irvine
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 1477
Record Dates: First submitted 2022-11-30; First posted 2022-12-21 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Blood Sugar; High; Blood Pressure; Dietary Habits
MeSH Terms: conditions — Hyperglycemia; Feeding Behavior | interventions — Microscopy, Electron, Scanning Transmission

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants are aware of study arm, but measured primary preliminary outcome is from a blinded CGM. Additionally, participants are not provided any of measured data during participation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Regular sweetened commercial foods (processed and high added sugar) (Experimental): This is the "usual" habits period. Participants consume the chosen, sweetened commercial products of their choice in the breakfast cereal/cereal-granola bar category (at least 1 daily serving) and sweetened baked goods/candy/desserts (at least 1 daily serving).
  * If they eat peanuts or nuts, and willingly consume chocolate covered peanuts or nuts, they will eat regular sweetened chocolate covered nuts/peanuts at least 3 days a week (1 serving/day), or as frequently as their usual habits if more often.
  * If they consume sweetened beverages (artificial or regular) or sweetened coffee or tea, they will consume these regular sweetened beverages as they usually do.
  Interventions: Other: Regular sweetened commercial foods
- Allulose sweetened commercial foods (processed and low added sugar) (Experimental): This period emphasizes minimizing added sugar, aligning intake levels with recommendations from the AHA and Dietary guidelines by consuming allulose sweetened products.
  Participants will eat at least 1 daily serving of the chosen, provided allulose sweetened breakfast/cereal-granola bar, and at least 1 daily serving of allulose sweetened baked goods/candy/desserts in place of the usual sweetened products from these food categories.
  * If they eat peanuts or nuts, and willingly consume chocolate covered peanuts or nuts, eat allulose sweetened chocolate covered nuts/peanuts at least 3 days a week (1 serving/day), or as frequently as usual habits if more often.
  * If they consume sweetened beverages (artificial or regular) or sweetened coffee or tea, consume allulose sweetened beverages in place of their artificial or regular sweetened beverages (provided commercial and/or syrups), and sweeten coffee or tea with the provided allulose sweetener. Do this according to usual habits.
  Interventions: Other: Allulose sweetened commercial foods
- Whole and minimally processed and sweetened foods (low processed and low added sugar) (Experimental): This period emphasizes incorporating minimally processed (e.g., intact whole grains) foods with minimal to no added sugar, aligning added sugar intake levels with recommendations from the American Heart Association and Dietary guidelines.
  Consume at least 1 daily serving of the chosen, minimal to no sweetened breakfast food in place of "usual" sweetened breakfast cereal/cereal-granola bar and consume a whole piece of fruit (or serving of fruit) in place of a sweetened baked goods/candy/desserts (at least 1 daily serving).
  * If they eat peanuts or nuts, consume plain or dry-roasted (no to low sodium) nuts/peanuts at least 3 days a week (1 serving), or as frequently as usual habits if more often
  * If consume sweetened beverages (artificial or regular) or sweetened coffee or tea, consume unsweetened coffee or tea and consume plain water in place of the sweetened beverages at the same frequency/amount that usually do
  Interventions: Other: Whole and minimally processed and sweetened foods

INTERVENTIONS:
Other: Regular sweetened commercial foods — This is your "usual" habits period. Consume the chosen, sweetened commercial products of your choice in the breakfast cereal/cereal-granola bar category (at least 1 daily serving) and sweetened baked goods/candy/desserts (at least 1 daily serving).
  * If you eat peanuts or nuts, and willingly consume chocolate covered peanuts or nuts, eat the regular sweetened chocolate covered nuts/peanuts at least 3 days a week (1 serving/day), or as frequently as your usual habits if more often.
  * If you consume sweetened beverages (artificial or regular) or sweetened coffee or tea, consume these regular sweetened beverages as you usually do.
  Other Names: Processed and high added sugar
  Arms: Regular sweetened commercial foods (processed and high added sugar)
Other: Allulose sweetened commercial foods — This period emphasizes minimizing added sugar, aligning intake levels with recommendations from the AHA and Dietary guidelines by consuming allulose sweetened products.
  Participants will eat at least 1 daily serving of the chosen, provided allulose sweetened breakfast/cereal-granola bar, and at least 1 daily serving of allulose sweetened baked goods/candy/desserts in place of the usual sweetened products from these food categories.
  * If they eat peanuts or nuts, and willingly consume chocolate covered peanuts or nuts, eat allulose sweetened chocolate covered nuts/peanuts at least 3 days a week (1 serving/day), or as frequently as usual habits if more often.
  * If they consume sweetened beverages (artificial or regular) or sweetened coffee or tea, consume allulose sweetened beverages in place of their artificial or regular sweetened beverages (provided commercial and/or syrups), and sweeten coffee or tea with the provided allulose sweetener. Do this according to usual habits.
  Other Names: Processed and low added sugar
  Arms: Allulose sweetened commercial foods (processed and low added sugar)
Other: Whole and minimally processed and sweetened foods — Consume at least 1 daily serving of the chosen, minimal to no sweetened breakfast product in place of your "usual" sweetened breakfast cereal/cereal-granola bar and consume a whole piece of fruit (or serving of fruit) in place of a sweetened baked goods/candy/desserts (at least 1 daily serving).
  * If you eat peanuts or nuts, consume plain or dry-roasted (no to low sodium) nuts/peanuts at least 3 days a week (1 serving), or as frequently as your usual habits if more often
  * If you consume sweetened beverages (artificial or regular) or sweetened coffee or tea, consume unsweetened coffee or tea and consume plain water in place of the sweetened beverages at the same frequency/amount that you usually do.
  This period emphasizes incorporating minimally processed (e.g., intact whole grains) foods with minimal to no added sugar, aligning added sugar intake levels with recommendations from the American Heart Association and Dietary guidelines.
  Other Names: Low processed and low added sugar
  Arms: Whole and minimally processed and sweetened foods (low processed and low added sugar)

SUMMARY:
The average adult in the US consumes over 1/3 of a cup of sugar each day, or nearly 300 calories worth, with the primary sources being from beverages, desserts and sweet snacks, candy, additions to beverages, and foods such as breakfast cereals. This is a risky health behavior, as high added sugar intake relates to higher risk of gaining weight, blood sugar disorders such as type 2 diabetes, plus heart disease and various cancers. Thus, high added sugar intake is problematic, and something in need of reducing. Therefore, the investigators are proposing to test how commercial foods sweetened with a new, FDA approved rare sugar with net zero calories (allulose), that is derived from dried fruits, brown sugar, and maple syrup may impact added sugar intake and usual blood sugar levels. The investigators are doing this by a randomized trial, in which the investigators will recruit participants with abnormal blood sugars (prediabetes or diabetes) or higher metabolic risk (bigger waist and elevated blood pressure or blood cholesterol) and ask them in random order to include foods in their usual dietary intake that are sweetened by regular sugars (regular sugar), foods that are sweetened by the zero calorie rare sugar allulose (low added sugar), or low added sugar intake by higher intake of fresh fruits and minimally processed and sweetened foods in place of usual sweetened foods. The investigators will measure their usual blood sugar levels for each of these 3 different 2- week periods with a blood glucose monitor, along with what they eat each of those periods, their blood pressure, and how the different dietary approaches impact how they feel.

DETAILED DESCRIPTION:
The average adult in the United States consumes around 17 teaspoons a day of added sugar, or nearly 280 calories, far exceeding recommended levels; and the leading sources of added sugars in the US diet are sugar-sweetened beverages, desserts and sweet snacks, candy, additions to coffee and teas, and substantial but insidious levels in foods such as brefakfast cereals. Indeed, this is fueled by intake of ultra-processed foods, which provide 58 % of energy intake and 89 % of added sugars in the American diet. A significant body of evidence links high intake of added sugars to the spectrum of chronic diseases which predominate the current, era, particularly those impacted by glycemia, and particularly postprandial glycemia, which has a clear role in health and disease. Thus, it is no surprise that a leading health indicator for Healthy People 2030 is to "reduce consumption of added sugars by people aged 2 years and over". Despite myriad efforts to reduce sugar-sweetened beverage intake (which has occurred on some levels), levels of added sugars have continued to increase over the past decade. A major bottleneck in addressing the goal of reducing added sugars in the American diet has been the lack of products lower in added sugars or sugar-free that the average adult in the US finds palatable and doesn't carry ingrained stigma or taste preferences which limit intake (i.e., sweetened by FDA approved artificial sweeteners). Very recently, a potential solution to this bottleneck has appeared in the form of allulose, a natural "zero calorie" sweetener found in small amounts of maple syrup, dried fruits, and brown sugar. This sweetener is intended to be incorporated into bakery products, beverages, confectionaries, dairy products and as a straight sugar substitute. Additionally, there is preliminary evidence from basic science, and small trials in humans that shows benefit of intake in place of regular added sugar in both healthy populations and in individuals with type 2 diabetes in respect to glycemic dynamics. Thus, there is a need to begin testing whether intake of commercial products sweetened with allulose can indeed be an approach to reduce added sugar intake and improve glycemia, particularly in people with metabolic abnormalities who are more sensitive to added sugar intake.

Therefore, the investigators are proposing the following specific aims for this pilot study.

Aim 1: To inform hypotheses and test the preliminary effectiveness of the ability of commercial products sweetened with allulose to reduce added sugar intake and reduce measures of glycemia, the investigators will carry out a randomized crossover dietary intervention with provision of categories of participant chosen food with specific consumption instructions, that compares a period of intake of regular sweetened commercial foods (processed and high added sugar), a period of intake of allulose sweetened commercial products (processed and low added sugar), and a period emphasizing whole and minimally processed and sweetened foods (low processed and low added sugar).

Aim 2: The investigators will measure dietary intake to estimate diet quality in each period, as well as measure blood pressure, weight, and psychosocial measures to provide a comprehensive initial impact of these approaches, and inform hypotheses for longer and more comprehensive future research.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes with HbA1c < 8.5%, or prediabetes (defined by HbA1c of 5.7-6.4%) or fasting glucose (≥ 100 mg/dl )
* or abdominal obesity (defined by sex and ethnic based thresholds: Europid/Sub-Saharan Africa/E Med-Middle E ethnicity (M 94 cm / F 90 cm), S/SE/E Asian and ethnic S and Central Americans (M 90 cm / F 80 cm) with at least one other abnormality from the following: (elevated triglycerides (≥ 150 mg/dl), elevated LDL (≥ 130 mg/dl or Rx), low HDL (<40 mg/dl M, <50 mg/dl F, or Rx), elevated blood pressure (>130 systolic or > 85 diastolic, or Rx).
* Free of clinically significant or unstable pulmonary, cardiovascular, gastrointestinal, hepatic, or renal functional abnormality; or currently pregnant.
* Weight stable for past 3 months (+- 5% of current body weight) and not planning to lose or gain weight over study period.
* able to provide informed consent
* otherwise healthy (beyond above noted health criteria), who meet the following criteria: interested in participating in and adhering to the prescribed 6-week long study comprised of 3, 2-week periods
* access to a telephone
* a stable dietary history, defined as neither introducing nor eliminating a major food group in their diet for at least the previous month
* eat a breakfast meal or morning snack (defined as an eating occasion after waking and before eating a lunch meal) 5 or more times a week on average
* 2 servings a day of food/beverage with > 20% of added sugar intake for day (10 g/serving) as estimated from dietary and beverage survey

Exclusion Criteria:

* Never diagnosed with Alzheimer's disease or related dementias, or any cognitive related conditions (interfere with ability to participate and respond to outcome assessments)
* Currently pregnant (self-report) or planning to become pregnant during study period, -Current participation in another interventional clinical trial
* Previous randomization in the study
* Current treatment for cancer
* Systolic blood pressure >160 mm Hg or diastolic blood pressure >100 mm Hg
* Major surgery planned during study duration
* Any disease or health condition which requires adherence to a specific diet/eating pattern that would prohibit participation
* Food insecurity assessed by Six-Item Short Form of the Food Security Survey Module (score > 1)
* Not responsible for choice of > 50% of dietary intake,
* work or obligations that require being awake during 3rd or overnight shift
* > 14 alcohol drinks /week
* heavy marijuana/THC product usage (> 5 days / week)

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2023-04-19 (Actual)

PRIMARY OUTCOMES:
Glycemic Variability (and specifically the Coefficient of Variation -CV) | 14 days (each period)
  Measured via Blinded Continuous Glucose Monitoring (CGM). We will collect CGM data over the course of the study during each of the three, 14-day periods as the primary clinical measure. This is an apt measure that is meaningful and interpretable across the spectrum of glycemic/metabolic abnormality to frank type 2 diabetes. The inherent major influence of CV is postprandial glucose, which is meaningful across the same spectrum for disease risk. We will use the Abbott Freestyle Libre Pro system.

SECONDARY OUTCOMES:
CGM Time in Range | 14 days (each period)
  the amount of time spent in the target blood glucose (blood sugar) range-between 70 and 180 mg/dL
CGM Mean glucose | 14 days (each period)
  Mean glucose (mg/dL)
Blood pressure | End of each 14-day period
  Systolic and Diastolic blood pressure, standard clinical measurement
Dietary Quality | Each 14-day period
  HEI dietary quality score as derived from 3 unannounced 24-hour dietary recalls each period (1 weekend, 2 non-consecutive weekdays), scored 0-100, higher = better diet quality
Weight (kg) | End of each 14-day period
  Weight measured on standardized scale
Physical activity | 7-days Each period
  Mean MET/hour objective measured via Activpal
Sleep | 7-days Each period
  Mean hours/day Objectively measured via Activpal
Food preference and food reward | End of each 14-day period
  Leeds Food Preference Questionnaire
Quality of life and well-being (Short-Form 12, SF-12) | End of each 14-day period
  SF-12 The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality of life measure. with a range from 0 to 100, with higher scores representing better self-reported health

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Irvine, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: Undecided